CLINICAL TRIAL: NCT00288041
Title: A Phase II Trial of PS-341 in Combination With Paclitaxel and Carboplatin for the Treatment of Metastatic Melanoma
Brief Title: Bortezomib, Paclitaxel, and Carboplatin in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00138; MC047C; N01CM62205 (NIH)
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Ciliary Body and Choroid Melanoma, Medium/Large Size; Extraocular Extension Melanoma; Iris Melanoma; Recurrent Intraocular Melanoma; Recurrent Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — Carboplatin; Paclitaxel; Taxes; Bortezomib

ARMS (1):
- Treatment (bortezomib, paclitaxel, carboplatin) (Experimental): Patients will receive an infusion of bortezomib twice in week 1 and once in week 2. They will also receive a 3-hour infusion of paclitaxel and an infusion of carboplatin once in week 1. Treatment may repeat every 3 weeks for as long as benefit is shown.
  Interventions: Drug: carboplatin; Drug: paclitaxel; Drug: bortezomib

INTERVENTIONS:
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE

SUMMARY:
This phase II trial is studying how well giving bortezomib together with paclitaxel and carboplatin works in treating patients with metastatic melanoma. Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Bortezomib may help paclitaxel and carboplatin kill more tumor cells by making tumor cells more sensitive to these drugs

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the confirmed tumor response rate and adverse event profile of bortezomib, carboplatin, and paclitaxel as first-line therapy for patients with metastatic melanoma.

SECONDARY OBJECTIVE:

I. Evaluate time to tumor progression, overall survival, and duration of response.

OUTLINE: This is a multicenter study.

Patients receive bortezomib intravenously (IV) over 3-5 seconds on days 1, 4, and 8 and paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 2. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 3 years.

ELIGIBILITY:
Criteria:

* No uncontrolled intercurrent illness including any of the following: ongoing or active infection; symptomatic congestive heart failure; unstable angina pectoris; cardiac arrhythmia
* No psychiatric illness that would limit compliance with study requirements
* No other uncontrolled serious medical conditions (e.g., diabetes)
* No more than 1 prior cytotoxic chemotherapy regimen
* No more than 2 prior immunotherapy regimens either in adjuvant or metastatic setting
* At least 4 weeks since prior major radiotherapy or chemotherapy
* At least 8 weeks since prior monoclonal antibody therapy
* At least 4 weeks since prior immunotherapy or biologic therapy
* At least 3 weeks since prior surgery
* Recovered from prior therapies
* No prior therapy with bortezomib, paclitaxel, or carboplatin
* No other prior or concurrent chemotherapy, immunotherapy, radiotherapy, or any other therapy or supportive care considered investigational
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent prophylactic colony-stimulating factors
* Histologically confirmed malignant melanoma
* Patients with significant fluid retention, including ascites or pleural effusion, may be allowed at the discretion of the principal investigator
* No known brain metastases by brain imaging with contrast
* Absolute neutrophil count >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Routine urine analysis with predicted 24-hour urine protein < 500 mg OR 1+ proteinuria by urine dipstick with 24-hour urine protein < 500 mg
* Total bilirubin < 1.5 mg/dL
* AST =< 3 times ULN
* Creatinine =< 1.5 times ULN
* ECOG performance status (PS) 0, 1, or 2 (Karnofsky PS >= 60%)
* Life expectancy by physician estimate > 12 weeks
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 6 months after completion of study treatment
* Negative pregnancy test
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to bortezomib
* No peripheral neuropathy >= grade 2
* Manifestations of stage IV disease (e.g., cutaneous, uveal)
* All melanomas, regardless of origin, allowed
* Measurable disease, defined as at least one lesion whose longest diameter can be accurately measured as >= 2.0 cm with conventional techniques or as >= 1.0 cm with spiral CT scan
* No nonmeasurable disease only, including any of the following: bone lesions, leptomeningeal disease, ascites, pleural/pericardial effusion, inflammatory breast disease, lymphangitis cutis/pulmonis, abdominal masses that are not confirmed and followed by imaging techniques, cystic lesions
* Hemoglobin >= 9.0 g/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2005-10; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Confirmed tumor response rate defined as the total number of evaluable patients whose objective tumor status is either a complete or partial response according to the RECIST criteria | Assessed up to 3 years
  If at most 3 of the first 19 eligible patients enrolled achieved a partial or complete response by the RECIST criteria, then enrollment would be terminated and the regimen would be considered inactive in this patient population. A 90% confidence interval will be constructed using the Duffy-Santer approach.
Adverse event profile as measured by NCI-CAE version 3.0 | Assessed up to 3 years
  The maximum grade for each type of toxicity will be recorded for each patient at each evaluation. The frequency and severity of each type of toxicity will be determined overall and by course.

SECONDARY OUTCOMES:
Time to disease progression | From registration to documentation of disease progression, assessed up to 3 years
  Estimated using the Kaplan-Meier method.
Duration of response | From the date at which the patient's objective status is first noted to be either a CR or PR to the date progression is documented, assessed up to 3 years
  Estimated using the Kaplan-Meier method.
Survival time | From registration to death due to any cause, assessed up to 3 years
  Estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Croghan, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States